CLINICAL TRIAL: NCT03906266
Title: Comparison of the Efficacy of Adductor Pollicis, NRS 2002, Nutric and SGD Tests in Assessing Nutritional Status in Patients With Sepsis
Brief Title: Assessing Nutritional Status in Patients With Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Prof Mehmet Turan Inal, Principal Investigator, Clinical Professor, Trakya University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: TÜTF-BAEK 2016/146
Record Dates: First submitted 2018-12-17; First posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: tests for understanding nutritional deficiency will be compared in a single patient group
Who Masked: Investigator
Masking Description: tests are made by different persons
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- nutric score (Active Comparator): > 5 indicates high risk for malnutrition < 4 indicates low risk for malnutrition
  Interventions: Diagnostic Test: NRS 2002, nutric, SGA and adductor pollicis
- adductor pollicis (Placebo Comparator): < 20 mm indicates high high risk for malnutrition > 20 mm indicates low risk for malnutrition
  Interventions: Diagnostic Test: NRS 2002, nutric, SGA and adductor pollicis
- SGA score (Placebo Comparator): SGA 1 indicates no malnutrition SGA 2 indicates good diet SGA 3 indicates high risk for malnutrition
  Interventions: Diagnostic Test: NRS 2002, nutric, SGA and adductor pollicis
- NRS 2002 score (Placebo Comparator): > 3 indicates high risk for malnutrition
  Interventions: Diagnostic Test: NRS 2002, nutric, SGA and adductor pollicis

INTERVENTIONS:
Diagnostic Test: NRS 2002, nutric, SGA and adductor pollicis — NRS 2002, nutric, SGA and adductor pollicis tests detects the malnutrition

SUMMARY:
In this study, the investigators aimed to investigate the efficacy of NRS-2002, SGA, nutric and adductor pollicis longus muscle thickness tests in patients with sepsis in intensive care unit. The patients will be diagnosed with sepsis according to 2013 sepsis diagnostic criteria. In these diagnostic criteria, the systemic inflammatory reaction syndrome criteria are fever> 38.3 ° C or <36 ° C,> 12000 / mm3 or <4000 / mm3, or more than 10% banded leucocytes, the respiratory rate is greater than 20 / min or In case of two suspected outbreaks> 90 / min., or suspected infection or culture-proven infection, the patient will be diagnosed with sepsis.

NRS-2002, nutric and SGA tests will be performed in all patients who are diagnosed with sepsis and are expected to stay in intensive care for more than 24 hours. Adductor pollicis longus muscle thickness will be measured in the same patients to understand the effectiveness of these tests on malnutrition. All tests are painless procedures. Adductor pollicis longus muscle measuring apparatus is available in intensive care.

DETAILED DESCRIPTION:
The majority of patients in the intensive care unit are diagnosed with sepsis. Malnutrition is frequently observed in these patients, and malnutrition can be detected by tests performed in patients such as NRS-2002, nutric and SGA. The parameters evaluated in the SGA test are: the investigatorsight loss in the last 6 months, the investigatorsight loss in the last 2 the investigatorseks, changes in oral intake, dietary changes, nausea, vomiting, diarrhea, functional capacity, subcutaneous fat evaluation, muscle loss assessment, edema and acid. All these parameters are evaluated with the help of a scale and the patient's malnutrition status is classified as A, B, C. Group A is mild, group B is medium and group C indicates heavy malnutrition. This test is a test that can be carried out at bedside. In the other test, NRS-2002, the patient is scored according to the patient's nutritional status and the severity of the disease. Here, the score is greater than ≥3 indicates that the patient is at risk of malnutrition. <Less than 3 indicates that the patient should be screened once a the investigatorsek. In the measurement of adductor pollicis longus muscle thickness in recent years, adductor pollicis longus muscle thickness betthe investigatorsen the thumb and forefinger in the patient's dominant hand is measured. This value has been shown to be valuable in determining the malnutrition status of the studies.

In our study, the investigators aimed to investigate the efficacy of these three values in patients with sepsis in intensive care unit. The patients will be diagnosed with sepsis according to 2013 sepsis diagnostic criteria. In these diagnostic criteria, the systemic inflammatory reaction syndrome criteria are fever> 38.3 ° C or <36 ° C,> 12000 / mm3 or <4000 / mm3, or more than 10% banded leucocytes, the respiratory rate is greater than 20 / min or In case of two suspected outbreaks> 90 / min., or suspected infection or culture-proven infection, the patient will be diagnosed with sepsis.

NRS-2002, nutric and SGA tests will be performed in all patients who are diagnosed with sepsis and are expected to stay in intensive care for more than 24 hours. Adductor pollicis longus muscle thickness will be measured in the same patients to understand the effectiveness of these tests on malnutrition. These tests will be carried out only once. All tests are painless procedures. Adductor pollicis longus muscle measuring apparatus is available in intensive care.

ELIGIBILITY:
Inclusion Criteria:

patients in the ICU for more than 24 hours patients with sepsis

Exclusion Criteria:

under 18 years old over 90 years old patients who dot have sepsis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
to understand the best malnutrition screening test | 18 months
  Our aim was to access which malnutrition test was the best

IPD SHARING:
Plan to Share IPD: No